CLINICAL TRIAL: NCT07154316
Title: A Randomized Phase II Study of Long-term Chemoradiotherapy or Short-term Radiotherapy Combined With CAPOX, PD-1 Monoclonal Antibody and COX-2 Inhibitors in MSS Type Locally Advanced Rectal Cancer
Brief Title: Phase II RCT of LCRT vs SCRT + CAPOX/PD-1i/COX-2i in MSS Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Anyang Tumor Hospital (Other); Fujian Cancer Hospital (Other Government); Shandong First Medical University (Other); Yunnan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Li Dawei, PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SERRAC
Record Dates: First submitted 2025-07-30; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-course chemoradiotherapy group (Experimental): The long-course chemoradiotherapy (LC-CRT) arm refers to a preoperative treatment regimen combining normofractionated radiotherapy with concurrent chemotherapy.
  Interventions: Radiation: LCRT; Drug: CAPOX; Drug: PD-1; Drug: Celecoxib
- Short-course chemoradiotherapy group (Experimental): The short-course chemoradiotherapy group refers to a preoperative regimen combining hypofractionated radiotherapy with concurrent or sequential chemotherapy .
  Interventions: Radiation: SCRT; Drug: CAPOX; Drug: PD-1; Drug: Celecoxib

INTERVENTIONS:
Radiation: LCRT — 50Gy/25Fx
  Arms: Long-course chemoradiotherapy group
Radiation: SCRT — 25Gy/5Fx
  Arms: Short-course chemoradiotherapy group
Drug: CAPOX — 1000mg/m2 bid d1-14
Drug: PD-1 — 300mg d1，q3w
Drug: Celecoxib — 200mg, bid

SUMMARY:
This randomized phase II trial evaluates the efficacy of long-course chemoradiotherapy (50Gy/25Fx + capecitabine) versus short-course radiotherapy (25Gy/5Fx) combined with CAPOX（Capecitabine and Oxaliplatin）, PD-1 inhibitor (serplulimab), and COX-2 inhibitor (celecoxib) in MSS（MicroSatellite Stable） locally advanced rectal cancer, with primary endpoint of complete response rate (pCR+cCR)（Complete Remission） and secondary endpoints including anal preservation rate and 3-year survival outcomes, aiming to elucidate the immunomodulatory effects of triple therapy on tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, regardless of gender.
* Pathologically confirmed rectal adenocarcinoma.
* Tumor located ≤10 cm from the anal verge.
* Baseline stage T3-4 and/or N+ (locally advanced disease).
* No evidence of distant metastasis.
* Microsatellite stability (MSS) or proficient mismatch repair (pMMR).
* Karnofsky Performance Status (KPS) ≥70.
* No prior chemotherapy or any other anticancer therapy before enrollment.
* No prior immunotherapy.
* Able to comply with study protocol requirements throughout the study period.
* Signed written informed consent obtained prior to study participation.

Exclusion Criteria:

* Pregnant or lactating women.
* Individuals with a history of other malignant diseases within the past 5 years, excluding cured skin cancer and cervical carcinoma in situ.
* Individuals with a history of uncontrolled epilepsy, central nervous system diseases, or mental disorders, where the clinical severity (as judged by the investigator) may impair the ability to sign the informed consent form or affect compliance with oral medication.
* Clinically significant (i.e., active) heart disease, including symptomatic coronary heart disease, congestive heart failure of New York Heart Association (NYHA) class II or worse, severe arrhythmias requiring pharmacological intervention, or a history of myocardial infarction within the past 12 months.
* Individuals requiring immunosuppressive therapy for organ transplantation and those on long-term corticosteroid therapy.
* Individuals with autoimmune diseases.
* Individuals with severe, uncontrolled, recurrent infections or other severe, uncontrolled concurrent diseases.
* Baseline blood routine and biochemical parameters not meeting the following criteria: hemoglobin ≥90 g/L; absolute neutrophil count (ANC) ≥1.5×10⁹/L; platelets ≥100×10⁹/L; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× upper limit of normal (ULN); alkaline phosphatase (ALP) ≤2.5×ULN; serum total bilirubin <1.5×ULN; serum creatinine <1×ULN; serum albumin ≥30 g/L.
* Individuals with known dihydropyrimidine dehydrogenase (DPD) deficiency. Individuals with a history of hypersensitivity to any component of the study medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
CR (Complete Response) | 3 years
  Complete response (CR) in malignant tumor patients is defined as the complete disappearance of all target lesions, normalization of tumor marker levels, and absence of new lesions for ≥4 weeks after treatment.

SECONDARY OUTCOMES:
sphincter preservation rate | 3 years
Grade 3 or higher toxicity rate | 3 years
3yPFS (Progression-Free Survival) | 3 years
  PFS (Progression-Free Survival) in oncology is defined as the time from the initiation of treatment to the occurrence of disease progression or death from any cause , whichever occurs first.
3yLRFS (Local Recurrence-Free Survival) | 3 years
  LRFS (Local Recurrence-Free Survival) is a clinical endpoint in oncology that measures the time from treatment initiation to the occurrence of local recurrence or death from any cause , whichever occurs first, commonly used to assess tumor control efficacy after surgery or radiotherapy.
3yOS (Overall Survival) | 3 years
  Measures the time until death , regardless of cause, reflecting the ultimate therapeutic outcome .
Surgical complications | 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Yunnan Cancer Hospital, Kunming
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No